CLINICAL TRIAL: NCT06038370
Title: Self-induced Cognitive Trance to Improve Quality of Life of Patients With Chronic
Brief Title: Self-induced Cognitive Trance for Chronic Pain Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Audrey Vanhaudenhuyse, Head, University of Liege
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-85
Record Dates: First submitted 2023-08-29; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Chronic Pain
Keywords: Self-induced cognitive trance; Non-ordinary state of consciousness; Pain; Quality of life
MeSH Terms: conditions — Chronic Pain; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self-induced cognitive trance (Experimental)
  Interventions: Behavioral: Self-induced cognitive trance

INTERVENTIONS:
Behavioral: Self-induced cognitive trance — The cognitive trance-based intervention will consist of a two-day workshop in groups of approximately 10 participants, where they will learn how to induce the cognitive trance, with the use of different sound-loops that can induce trance in untrained people in a safe way. After two weeks of home practice, participants will redo a two-day consolidation training. At-home practice is encouraged between sessions.

SUMMARY:
The need to find complementary approaches, based on a holistic perspective of the human being, takes on its full meaning in a political context that recommends efficient health programs. Self-induced cognitive trance is one of these complementary approaches, which induce a non-ordinary state of consciousness. The aim of this work is to evaluate whether learning self-induced cognitive trance can improve the quality of life of people with chronic pain. Participants will participate in two times two days workshop aiming at learning how to self-induce cognitive trance. Pain, Fatigue, anxiety, depression, attitudes towards pain, and quality of life will be assessed before and after each workshops. Two follow-ups at 6 and 12 months afer the last workshop will be caried out were outomes will be assessed. Furthmore, questionnaires related to the phenomenology of self-induced cognitive trance will be adeministrered. Investigators also proceeded to interveiwes after the second workshop to gather qualitative information.

ELIGIBILITY:
Inclusion Criteria:

* French speacking
* Chronic pain
* On stable pharmacological treatment over the last four months

Exclusion Criteria:

* Psychiatric disorders,
* drug addiction
* alcoholism

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2024-02-10 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Assessed before the intervention, immediately after the first workshop, immediately after the second workshop and at 6- and 12-month follow-up
  Visual Analog Scale will be used to assess pain, at the present moment, at its weakest and strongest, on a scale of 0 (no pain) to 10 (worst pain imaginable)
Fatigue intensity | Assessed before the intervention, immediately after the first workshop, immediately after the second workshop and at 6- and 12-month follow-up
  Visual Analog Scale will be used to assess pain, at the present moment, at its weakest and strongest, on a scale of 0 (no pain) to 10 (worst pain imaginable)
Anxiety | Assessed before the intervention, immediately after the first workshop, immediately after the second workshop and at 6- and 12-month follow-up
  Hospital Anxiety and Depression scale comprises 14 items subdivided into 7 sub-items, each linked to a subscale, one for the level of anxiety and one for the level of depression, for a total score ranging from 0 to 21 for each of these subscales. A score of 0 to 7 is equivalent to a "normal" state, a score of 8 to 10 suggests only the presence of a mood disorder, a score of 11 to 15 indicates the probable presence of a moderate mood disorder, and finally, a score above 16 indicates a severe mood disorder.
Depression | Assessed before the intervention, immediately after the first workshop, immediately after the second workshop and at 6- and 12-month follow-up
  Hospital Anxiety and Depression scale comprises 14 items subdivided into 7 sub-items, each linked to a subscale, one for the level of anxiety and one for the level of depression, for a total score ranging from 0 to 21 for each of these subscales. A score of 0 to 7 is equivalent to a "normal" state, a score of 8 to 10 suggests only the presence of a mood disorder, a score of 11 to 15 indicates the probable presence of a moderate mood disorder, and finally, a score above 16 indicates a severe mood disorder.
Attitudes towards pain | Assessed before the intervention, immediately after the first workshop, immediately after the second workshop and at 6- and 12-month follow-up
  The Survey of Pain Attitude-35. It is composed of 7 subscales: perceived disability measures the belief that disability is caused by pain; pain-injury link assesses the belief that pain is a physical injury; medication measures the belief that medication is the only remedy, solicitude measures the belief that those around patients should assist them in their painful experience, expectation of cure measures the belief that doctors are responsible for reducing their pain, perceived control assesses the feeling of perceived control, and finally, emotion measures the feeling that emotions have an impact on pain. Scores are specific to each scale. The higher the score, the more patients hold this belief.
Quality of life | Assessed before the intervention, immediately after the first workshop, immediately after the second workshop and at 6- and 12-month follow-up
  The Short From Health Survey assesses overall quality of life. It comprises 36 items subdivided into 9 subscales: physical functioning, limitations resulting from physical health, limitations resulting from emotional health, vitality (energy/fatigue), emotional well-being, social functioning, pain, general state of health and, finally, changes in state of health. Each of these scales is weighted by a score ranging from 0 to 100. The first 8 dimensions of the SF-36 are grouped into 2 synthetic scores. A physical score (PCS) groups the 8 dimensions according to a weighting that favors the physical component, while the mental score (MCS) summarizes the mental component of the dimension scores. The higher the scores, the better the mental and physical health. The final item assesses perceived change in health status.
Global Impression of change | Assessed before the intervention, immediately after the first workshop, immediately after the second workshop and at 6- and 12-month follow-up
  Global Impression of change assesses patients' beliefs about the effectiveness of their treatment on their disease. It's a simple scale that goes up to 7 points, equivalent to the best possible improvement.

SECONDARY OUTCOMES:
Positive affect | Assessed before the intervention, immediately after the first workshop, immediately after the second workshop and at 6- and 12-month follow-up
  The Positive Affect and Negative Affect Schedule is dedicated to measuring mood and feelings. The questionnaire comprises two scales. The first measures positive affect, the second negative affect. Each scale comprises 10 items, for a total of 20 items, and each item is rated on a scale from 1 (very little or not at all) to 5 (very much or not at all).
Negative affect | Assessed before the intervention, immediately after the first workshop, immediately after the second workshop and at 6- and 12-month follow-up
  The Positive Affect and Negative Affect Schedule is dedicated to measuring mood and feelings. The questionnaire comprises two scales. The first measures positive affect, the second negative affect. Each scale comprises 10 items, for a total of 20 items, and each item is rated on a scale from 1 (very little or not at all) to 5 (very much or not at all).
Ego-Dissolution | Assessed before the intervention, immediately after the first workshop, immediately after the second workshop and at 6- and 12-month follow-up
  Ego-Dissolution Inventory comprises 16 items subdivided into 2 subscales representing ego inflation and ego dissolution, each scale comprising 8 items. Each item is monitored by a numerical score ranging from 0 (no, no more than usual) to 100 (yes, entirely or completely).
Mystical Experience | Assessed before the intervention, immediately after the first workshop, immediately after the second workshop and at 6- and 12-month follow-up
  Mystical Experiences Questionnaire comprises 30 items divided into 4 subscales representing mysticism, which qualifies experiences of communication with a reality that cannot be discerned by common sense, positive mood, transcendence of time and space, and ineffability, which represents the experience of being able to communicate with a reality that cannot be discerned by common sense. considers that the experience cannot be described in words, each item is evaluated with a score ranging from 0 (none, not at all) to 5 (extreme, more than any other moment in my life and more than 4).
Phenomenology of trance | Assessed before the intervention, immediately after the first workshop, immediately after the second workshop and at 6- and 12-month follow-up
  Assessed through a self-made questionnaire. It consists of 10 questions, each of which is evaluated by a score ranging from 1 (strongly disagree) to 7 (strongly agree).
Experience with trance | Immediately after the second workshop
  Semi-structured interview

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - CHU of Liège, Liège
  - University of Liège, Liège

IPD SHARING:
Plan to Share IPD: Undecided